CLINICAL TRIAL: NCT05355402
Title: A Randomized, Double-blind, Placebo-Controlled, Phase 2b Study of ISIS 678354 in Patients With Hypertriglyceridemia and Atherosclerotic Cardiovascular Disease (Established or at Increased Risk for), and/or With Severe Hypertriglyceridemia
Brief Title: A Study of Olezarsen (Formerly Known as AKCEA-APOCIII-LRx) in Adults With Hypertriglyceridemia and Atherosclerotic Cardiovascular Disease (Established or at Increased Risk for), and/or With Severe Hypertriglyceridemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ISIS 678354-CS8
Expanded Access: NCT06360237 (Approved for marketing)
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Hypertriglyceridemia; Atherosclerotic Cardiovascular Disease; Severe Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia; Atherosclerosis | interventions — olezarsen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Olezarsen (Experimental): Olezarsen will be administered once every 4 weeks by subcutaneous (SC) injection for up to 49 weeks.
  Interventions: Drug: Olezarsen
- Placebo (Placebo Comparator): Olezarsen-matching placebo will be administered once every 4 weeks by SC injection for up to 49 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Olezarsen — Olezarsen will be administered by SC injection.
  Other Names: ISIS 678354; AKCEA-APOCIII-LRx
  Arms: Olezarsen
Drug: Placebo — Olezarsen-matching placebo will be administered once every 4 weeks by SC injection for up to 49 weeks.
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the effect of olezarsen on percent change in fasting triglyceride (TG) levels compared to placebo at Months 6 and 12 and the percentage of participants who achieve different thresholds in fasting TG. Another objective is to evaluate the effect of olezarsen on percent change in fasting apolipoprotein C-III (apoC-III), very low-density lipoprotein cholesterol (VLDL-C), remnant cholesterol, non-high-density lipoprotein cholesterol (non-HDL-C), HDL-C, total cholesterol (TC), apolipoprotein B (apoB), low-density lipoprotein cholesterol (LDL-C), and apolipoprotein A-1 (apoA-1).

DETAILED DESCRIPTION:
This will be a multi-center, randomized, double-blind, placebo-controlled study in approximately 152 participants with hypertriglyceridemia (triglycerides > 150 milligrams per deciliter [mg/dL]) and established or at increased risk for atherosclerotic cardiovascular disease, and/or with severe hypertriglyceridemia. The study will have an up to 8-week screening period, a 53-week treatment period, and a 13-week post-treatment follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years at the time of informed consent
2. Fall into at least 1 of the following groups (a or b):

   1. Hypertriglyceridemia with fasting TG ≥ 150 mg/dL (1.69 millimoles per liter [mmol/L]) and < 500 mg/dL (5.65 mmol/L) with either clinical diagnosis of atherosclerotic cardiovascular disease (ASCVD) or at increased risk for ASCVD
   2. Severe hypertriglyceridemia with fasting TG ≥ 500 mg/dL (5.65 mmol/L).
3. Participants must be on standard-of-care (SOC), lipid-lowering medications per local guidelines.
4. Participants must be willing to comply with diet and lifestyle recommendations as able.

Exclusion Criteria:

1. Diabetes with any of the following:

   1. Newly diagnosed within 12 weeks of screening
   2. Hemoglobin A1C (HbA1c) ≥ 9.5% at Screening
   3. Change in basal insulin regimen > 20% within 3 months prior to Screening
   4. For participants with type 1 diabetes: episode of diabetic ketoacidosis, or ≥ 3 episodes of severe hypoglycemia within 6 months prior to Screening
2. Acute coronary syndrome or stroke/transient ischemic attack (TIA) within 6 months prior to Screening
3. Major surgery, peripheral revascularization, or non-urgent percutaneous coronary intervention (PCI) within 3 months prior to Screening, or upcoming planned major surgery or major procedure (e.g., arterial revascularization) during the course of the study
4. Active pancreatitis within 4 weeks prior to Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Percent Change From Baseline at Month 6 (average of Weeks 25 and 27) in Fasting Triglycerides (TG) | Baseline and Month 6

SECONDARY OUTCOMES:
Percent Change From Baseline at Month 12 in Fasting TG | Baseline and Month 12
Proportion of Participants with Baseline TG < 500 mg/dL (5.65 mmol/L) Who Achieve Fasting TG < 150 milligrams per deciliter (mg/dL) (1.69 millimoles per liter [mmol/L]) at Month 6 | Baseline and Month 6
Proportion of Participants with Baseline TG < 500 mg/dL (5.65 mmol/L) Who Achieve Fasting TG < 150 mg/dL (1.69 mmol/L) at Month 12 | Baseline and Month 12
Proportion of Participants with Baseline TG ≥ 500 mg/dL Who Achieve Fasting TG < 500 mg/dL (5.65 mmol/L) at Month 6 | Baseline and Month 6
Proportion of Participants with Baseline TG ≥ 500 mg/dL Who Achieve Fasting TG < 500 mg/dL at Month 12 | Baseline and Month 12
Percent Change From Baseline at Months 6 and 12 in Fasting apoC-III | Baseline, Months 6 and 12
Percent Change From Baseline at Months 6 and 12 in Fasting VLDL-C | Baseline, Months 6 and 12
Percent Change From Baseline at Months 6 and 12 in Fasting Remnant Cholesterol | Baseline, Months 6 and 12
Percent Change From Baseline at Months 6 and 12 in Fasting Non-HDL-C | Baseline, Months 6 and 12
Percent Change From Baseline at Months 6 and 12 in Fasting HDL-C | Baseline, Months 6 and 12
Percent Change From Baseline at Months 6 and 12 in Fasting TC | Baseline, Months 6 and 12
Percent Change From Baseline at Months 6 and 12 in Fasting apoB | Baseline, Months 6 and 12
Percent Change From Baseline at Months 6 and 12 in Fasting LDL-C | Baseline, Months 6 and 12
Percent Change From Baseline at Months 6 and 12 in apoA-1 | Baseline, Months 6 and 12
Adjudicated acute pancreatitis event rate during the Treatment Period compared to placebo in patients with ≥ 2 events of adjudicated acute pancreatitis in 5 years prior to enrollment. | Baseline through Month 12
Adjudicated acute pancreatitis event rate during the Treatment Period compared to placebo. | Baseline through Month 12

CONTACTS AND LOCATIONS:
Locations (24):
- United States (21):
  - Clinical Trials Research, Lincoln, California
  - Catalina Research Institute, LLC, Montclair, California
  - Excel Medical Clinical Trials, LLC, Boca Raton, Florida
  - De La Cruz Research Center, Miami, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Research Physicians Network Alliance, Winter Park, Florida
  - IACT Health, Columbus, Georgia
  - Evanston Premier Healthcare Research, Evanston, Illinois
  - Clinical Investigation Specialist, Gurnee, Illinois
  - West Broadway Clinic, Council Bluffs, Iowa
  - Louisville Metabolic and Atherosclerosis Research Center (L-MARC), Louisville, Kentucky
  - Aa Mrc, Llc, Flint, Michigan
  - Clinical Research of South Nevada, Las Vegas, Nevada
  - Palm Research Center, Inc., Las Vegas, Nevada
  - Green and Seidner Family Practice Associates, Lansdale, Pennsylvania
  - Main Street Physicians Care Waterway, Little River, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - Tennessee Center for Clinical Trials, Tullahoma, Tennessee
  - Southern Endocrinology Associates, Mesquite, Texas
  - Manassas Clinical Research Center, Manassas, Virginia
  - York Clinical Research LLC, Norfolk, Virginia
- Canada (3):
  - Bluewater Clinical Research Group Inc, Sarnia, Ontario
  - Ecogene-21, Chicoutimi, Quebec
  - Clinique des Maladies Lipidiques de Quebec Inc., Québec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bergmark BA, Marston NA, Prohaska TA, Alexander VJ, Zimerman A, Moura FA, Murphy SA, Goodrich EL, Zhang S, Gaudet D, Karwatowska-Prokopczuk E, Tsimikas S, Giugliano RP, Sabatine MS; Bridge-TIMI 73a Investigators. Olezarsen for Hypertriglyceridemia in Patients at High Cardiovascular Risk. N Engl J Med. 2024 May 16;390(19):1770-1780. doi: 10.1056/NEJMoa2402309. Epub 2024 Apr 7. PMID 38587249